CLINICAL TRIAL: NCT05109572
Title: The Impact of the Covid-19 Pandemic on Schizophrenia Patients Registered With the Community Mental Health Center
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İsmail Koç, Specialist doctor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: 514/194/41
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Hospitalization; Emergency Medical Services

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hospitalized group: Hospitalized patient (HP) stayed in hospital during the Covid-19 pandemic period
  Interventions: Other: Non-hospitalized with emergency care; Other: Non-hospitalized and non-emergency care
- Non-hospitalized with Emergency care: Emergency care plan made but no hospitalization was included to this study during the Covid-19 pandemic period
  Interventions: Other: Hospitalized; Other: Non-hospitalized and non-emergency care
- Non-hospitalized and non-emergency care: Patients who neither apply to the emergency department nor are hospitalized was included to this study during the Covid-19 pandemic period
  Interventions: Other: Hospitalized

INTERVENTIONS:
Other: Hospitalized — It was developed by Addington et al. (1994) to measure the presence of depression and the severity of depressive symptoms in patients with schizophrenia. The scale consists of 9 items to assess depression and is answered with a four-point Likert scale. The validity and reliability of the scale in schizophrenia patients in the Turkish population was determined by Oksay et al. by (2000). In the reliability study, the Cronbach's alpha coefficient was found to be 0.88. The cut-off point of the scale was stated as 11.
  Groups: Non-hospitalized and non-emergency care; Non-hospitalized with Emergency care
Other: Non-hospitalized with emergency care — It is adapted from the Buss-Durkee Hostility Inventory by Buss and Perry (1992), the scale consists of 29 items and five-point Likert types. The scale is physical and verbal aggression, hostility, and anger. Questions 9 and 16 on the scale are reverse scored. The score value on the scale varies in direct proportion to the aggression, that is, the higher the score, the higher the aggression. The Cronbach Alpha internal consistency coefficients of the original version of the scale is defined as; 0.89 for physical aggression, 0.85 for physical aggression, 0.72 for verbal aggression, 0.77 for hostility, 0.83 for anger subscale.
  Groups: Hospitalized group
Other: Non-hospitalized and non-emergency care — Developed by Cull and Gill (1989), it evaluates the probability of suicide in adolescents and adults. The Turkish validity and reliability of the scale were performed by Atlı et al (2009). The scale consists of 36 items and is answered as a four-point Likert-type scale as "never or rarely", "sometimes", "often" and "often or always".
  Groups: Hospitalized group; Non-hospitalized with Emergency care

SUMMARY:
This study aimed to examine the effect of the Covid-19 pandemic on schizophrenia patients registered to the Community Mental Health Center (CMHC) in terms of depression, suicide risk, and tendency to violence.

DETAILED DESCRIPTION:
The study was conducted on patients registered to the Ministry of Health Kartal Dr. Lütfi Kırdar City Hospital Adatepe Community Mental Health Center and was followed up regularly. It was carried out on 108 individuals who met the diagnosis of schizophrenia according to the DSM-V (American Psychiatric Association 2013) and met the inclusion criteria. Individuals who were respectively classified as hospitalized group (HG) during the Covid-19 pandemic period (n=39), non-hospitalized with emergency care group (NHECG) without hospitalization (n=37), and non-hospitalized with non-emergency care group (NHNECG) (n=32). Individuals who had been diagnosed with schizophrenia for at least two years, were not in the active phase of the disease, did not have organic mental disorders, did not have any other psychiatric diseases were included in the study. In the study, the Socio-Demographic Questionnaire, the Calgary Depression Scale in Schizophrenia (CDSS), the Buss-perry Aggression Questionnaire (BPAQ), and the Suicide Probability Scale (SPS) were used.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-65,
* receiving service from Kartal Dr. Lütfi Kırdar City Hospital Adatepe CMHC,
* having been diagnosed with schizophrenia for at least two years,
* not being in the active phase of the disease,
* not having an organic mental disorder,
* not having an additional psychiatric illness, and
* being literate

Exclusion Criteria:

* Individuals with cognitive and physical dysfunction,
* mental retardation, different psychiatric diseases that would prevent interview or testing, and
* those who did not consent to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: receiving service and having been diagnosed with schizophrenia for at least two years by psychiatry who works from Kartal Dr. Lütfi Kırdar City Hospital Adatepe CMHC
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Calgary Depression Scale in Schizophrenia | 6 months
  It was developed by Addington et al. (1994) to measure the presence of depression and the severity of depressive symptoms in patients with schizophrenia. 19 The scale consists of 9 items to assess depression and is answered with a four-point Likert scale.The validity and reliability of the scale in
  schizophrenia patients in the Turkish population was determined by Oksay et al. by (2000). In the reliability study, the Cronbach's alpha coefficient was found to be 0.88. The cut-off point of the scale was stated as 11.
Buss-perry Aggression Questionnaire | 6 months
  It is adapted from the Buss-Durkee Hostility Inventory by Buss and Perry (1992), the scale consists of 29 items and five-point Likert types. 21 The scale is physical and verbal aggression, hostility, and anger. Questions 9 and 16 on the scale are reverse scored. The score value on the scale varies in direct proportion to the aggression, that is, the higher the score, the higher the aggression. The Cronbach Alpha internal consistency coefficients of the original version of the scale is defined as; 0.89 for physical aggression, 0.85 for physical aggression, 0.72 for verbal aggression, 0.77 for hostility, 0.83 for anger subscale.
Suicide Probability Scale | 6 months
  Developed by Cull and Gill (1989), it evaluates the probability of suicide in adolescents and adults. The Turkish validity and reliability of the scale were performed by Atlı et al (2009). The scale consists of 36 items and is answered as a four-point Likert-type scale as "never or rarely", "sometimes", "often" and "often or always".

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lütfi Kırdar Şehir Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided